CLINICAL TRIAL: NCT03495947
Title: Evaluation of Results of the Application of High Flow Nasal Cannula to Prevent the Failure of Extubation
Brief Title: High Flow Nasal Cannula in Immediately Post Extubation
Acronym: HFNC
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Sponsor
Other Study IDs: 3027
Record Dates: First submitted 2018-03-28; First posted 2018-04-12 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Airway Extubation; Oxygen Inhalation Therapy
Keywords: High Flow Nasal Cannula (HFNC).; Mechanical ventilation; Extubation failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: high flow nasal cannula — 24 hours of continuous use in the immediate post-extubation period.

SUMMARY:
The aim of the study is to determine the incidence of failure of extubation in high-risk patients using High Flow Nasal Cannula (HFNC) to prevent such failure in the Intensive Care Unit. A prospective cohort study was performed. To all adult patients receiving invasive mechanical ventilation ≥ 48 hours and ready for scheduled extubation according to tolerance of spontaneous breathing trial, with at least one of the criteria for high-risk for extubation failure (age greater than 65 years, hypoxemic acute respiratory failure as a cause of invasive mechanical ventilation, > 1 spontaneous ventilation test failed consecutive, history of chronic heart failure, history of chronic obstructive pulmonary disease or PaCO2> 45 mmHg, body mass index >30 kg/m2, post-operative solid organ transplantation), HFNC is applied for 24 hours. Demographic variables and clinical and gasometric parameters at the end of the spontaneous breathing trial, at 60 minutes, at 6 and 24 hours after the start of HFNC are recorded.

DETAILED DESCRIPTION:
At the end of the successful spontaneous breathing trial, clinical and gasometric parameters will be recorded and extubation will be performed. HFNC is placed with a flow of 50 l / m (only the flow is reduced before intolerance, at 5 l / min but only up to 40 l / min). Inspiratory oxygen fraction (FiO2) initially at 1 and progressively decreases until pulse oximeter saturation (SpO2) ≥ 92% is achieved. Said configuration is maintained for 60 minutes. After this time, arterial blood samples are taken and clinical and gasometric parameters are recorded in the follow-up chart. Based on them, behavior to be followed is defined. If "Fault criteria" are presented, a higher ventilatory support will be initiated. If not, continue with HFNC for the next 23 hours without exception. In this period the initial flow is maintained (40 to 50 l / min) and the FiO2 is programmed according to the SpO2 objective (≥ 92%). At 6 o'clock a new clinical and gasometric evaluation and data loading is carried out. 24 hours after the start of HFNC, a blood gas sample is taken and clinical and gasometric parameters are recorded. Treatment with HFNC is only suspended if the "Failure criteria" or the "Interruption criteria" are met. In the presence of the "Failure Criteria" and prior to delivering a greater ventilatory support, the clinical and gasometric parameters are recorded in the spreadsheet.

The data of categorical variables will be presented as frequency and percentage, while in quantitative variables, after testing normality by Shapiro-Wilks test, they will be presented as mean and standard deviation or median and interquartile range depending on their distribution. For comparisons between groups, chi-square or Fisher tests will be used, depending on the frequency expected in discrete and categorical variables, and in the continuous T or Mann-Whitney tests, depending on the type of distribution and variance. To determine the factors of risk of failure to extubation, a logistic regression study will be carried out with a system of selection of variables by forward steps. The odds ratio and its 95% confidence intervals will be calculated. Variables that are significant in the univariate study (p value <0.2) will be included in the multiple logistic regression study.

ELIGIBILITY:
Inclusion criteria:

- All adult patients receiving invasive mechanical ventilation ≥48 hours and ready for scheduled extubation according to tolerance of spontaneous breathing trial, with at least one of the following criteria for high-risk for extubation failure:

* Age greater than 65 years.
* Hypoxemic acute respiratory failure as a cause of invasive mechanical ventilation.
* >1 spontaneous ventilation test failed consecutive.
* History of chronic heart failure.
* History of chronic obstructive pulmonary disease or PaCO2 >45 mmHg.
* Body mass index >30 kg/m2.
* Post-operative solid organ transplantation.

Exclusion criteria:

* Need for orotracheal intubation and invasive mechanical ventilation (IOT / AVMI) according to the decision of the attending physician.
* Deterioration of the state of consciousness determined by Kelly Matthay's Scale >3.
* Hemodynamic instability: systolic blood pressure (TAS) <90 mmHg or TAM <65 mmHg despite receiving fluids and/ or vasopressors.
* Neuromuscular disease
* Neurocritical pathology.
* Epistaxis
* Skull base fracture, or inability to fix the HFNC.
* History of obstructive sleep apnea-hypopnea syndrome with indication and use of nocturnal continuous positive pressure.
* Participation in another research protocol of HFNC.

Elimination criteria

. Directives before or after the onset of a disease that limits the therapeutic effort and indicates not to intubate or perform cardiopulmonary resuscitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients receiving invasive mechanical ventilation ≥48 hours and ready for scheduled extubation according to tolerance of spontaneous breathing trial.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-01-03 (Actual); Study Completion 2019-01-03 (Actual)

PRIMARY OUTCOMES:
Extubation failure | In the first 48 hours
  the need to discontinue treatment with HFNC to progress to invasive or non-invasive ventilatory support within 48 hours of extubation.

SECONDARY OUTCOMES:
Time to failure of extubation | In the first 48 hours
  the date and time of extubation and start of HFNC will be recorded as well as the date and time of discontinuation of HFNC to progress to another type of ventilatory support within 48 hours following extubation.
Reasons for extubation failure | In the first 48 hours
  the cause of extubation failure
Type of ventilatory support post-failure of extubation | In the first 48 hours
  the type of ventilatory support post-failure will be recorded. Non-invasive mechanical ventilatory. Intubation orotracheal and invasive mechanical ventilatory.
Average time of use the HFNC | Through study completion, an average of 1 year
  the total hours of use of HFNC will be recorded
Length of stay in the Intensive care unit | Through study completion, an average of 1 year
  the total number of days of stay in the Intensive care unit will be recorded.
Incidence of mortality in the Intensive care unit | Through study completion, an average of 1 year
  the relationship between the total number of patients requiring HFNC and those who died after being included in the study will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Paulina E Ezcurra, Lic, Principal Investigator; Maria S Venuti, Dr, Principal Investigator
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464